CLINICAL TRIAL: NCT00627705
Title: Double-blind , Randomized, Placebo Controlled Study of N-Acetyl Cysteine in Autism.
Brief Title: A Study of N-Acetyl Cysteine in Children With Autism
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Antonio Hardan, Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SU-02012008-995; 10142
Record Dates: First submitted 2008-02-22; First posted 2008-03-03 (Estimated); Results first posted 2017-05-18 (Actual); Last update posted 2017-05-18 (Actual); Status verified 2017-04

CONDITIONS: Autistic Disorder
MeSH Terms: conditions — Autistic Disorder | interventions — Acetylcysteine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- N-Acetyl Cysteine (Active Comparator): active compound N-Acetyl Cysteine
  Interventions: Drug: N-Acetyl Cysteine
- Sugar pill (Placebo Comparator): Placebo or sugar pill
  Interventions: Other: Placebo - sugar pill

INTERVENTIONS:
Drug: N-Acetyl Cysteine — Phase 1: Oral, 900 mg daily for 4 weeks Phase 2: Oral, 900 mg twice daily 4 weeks Phase 3: Oral, 900 mg three times daily for 4 weeks
  Entire intervention lasts for 12 weeks (drug administration is continuous).
  Other Names: NAC
  Arms: N-Acetyl Cysteine
Other: Placebo - sugar pill — Phase 1: Oral, 900 mg daily for 4 weeks Phase 2: Oral, 900 mg twice daily 4 weeks Phase 3: Oral, 900 mg three times daily for 4 weeks
  Entire intervention lasts for 12 weeks (drug administration is continuous).
  Other Names: Placebo
  Arms: Sugar pill

SUMMARY:
The purpose of the study is to test the tolerability and efficacy of N-Acetyl Cysteine (NAC) in children with Autism. NAC is a compound that increases the levels of Glutathione, the body's main antioxidant. Glutathione is a compound in the blood that is part of a natural defense system (the antioxidant system). Anti-oxidants protect the body from damage caused by internal toxins called "free radicals." It is possible that children with Autism tend to have lower levels of glutathione, an important compound in our bodies that helps combat the effects of toxic free radicals.

We hope that by studying the antioxidant system in more detail, we will increase our understanding of the reasons why people develop Autism so that we can design better ways to treat individuals with this condition. This study is meant to test the safety tolerability of NAC and its effectiveness in the treatment of behavioral difficulties in children with autism. It will also examine the possible benefit of this agent in improving the core deficits in autism such as social deficits.

ELIGIBILITY:
Inclusion Criteria:

1. Outpatients between 3.0 and 12.11 years of age inclusive
2. Males and females who are physically healthy
3. diagnosis of autism based Diagnostic and Statistical Manual (DSM-IV-TR) criteria, the Autism Diagnostic Interview-Revised, and expert clinical evaluation
4. Clinical Global Impression Severity rating of 4
5. Care provider who can reliably bring subject to clinic visits, can provide trustworthy ratings, and interacts with subject on a regular basis
6. Ability of subject to swallow the compound
7. Stable concomitant medications for at least 2 weeks
8. No planned changes in psychosocial interventions during the open-label N-Acetyl Cysteine trial

Exclusion Criteria:

1. DSM-IV-TR diagnosis of schizophrenia, schizoaffective disorder, or psychotic disorder not otherwise specified
2. Prior adequate trial of N-Acetyl Cysteine
3. Active medical problems: unstable seizures, significant physical illness (e.g., serious liver or renal pathology)
4. Pregnancy or sexually active females
5. Subjects taking antioxidant agents and glutathione prodrugs will be excluded from the study except if they have been off these compounds for at least 4 weeks

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 43 (Actual)
Dates: Start 2008-02; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Hardan, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Hardan AY, Fung LK, Libove RA, Obukhanych TV, Nair S, Herzenberg LA, Frazier TW, Tirouvanziam R. A randomized controlled pilot trial of oral N-acetylcysteine in children with autism. Biol Psychiatry. 2012 Jun 1;71(11):956-61. doi: 10.1016/j.biopsych.2012.01.014. Epub 2012 Feb 18. PMID 22342106

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment started in March 2009 and ended in September 2010. This study was conducted in the Autism & Developmental Disabilities Clinic in the Division of Child & Adolescent Psychiatry, Lucile Packard Children's Hospital at Stanford University.
Pre-assignment Details: Fifty-one potential subjects inquired about the study. Forty-three of the subjects signed a consent form. Seven subjects were excluded because they did not meet criteria for autistic disorder. Three subjects decided not to participate in the study before baseline measures were obtained. Thirty-three subjects were randomized in the study.
Groups:
- N-Acetyl Cysteine: active compound N-Acetyl Cysteine
  N-Acetyl Cysteine: Phase 1: Oral, 900 mg daily for 4 weeks Phase 2: Oral, 900 mg twice daily 4 weeks Phase 3: Oral, 900 mg three times daily for 4 weeks
  Entire intervention lasts for 12 weeks (drug administration is continuous).
- Sugar Pill: Placebo or sugar pill
  Placebo - sugar pill: Phase 1: Oral, 900 mg daily for 4 weeks Phase 2: Oral, 900 mg twice daily 4 weeks Phase 3: Oral, 900 mg three times daily for 4 weeks
  Entire intervention lasts for 12 weeks (drug administration is continuous).
Period: Overall Study
Arm/Group | N-Acetyl Cysteine | Sugar Pill
Started | 15 | 18
Completed | 13 | 12
Not Completed | 2 | 6
Not completed — Unwilling to take the compound (taste) | 1 | 3
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | N-Acetyl Cysteine | Sugar Pill | Total
Number analyzed (Participants) | 15 | 18 | 33
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 15 | 18 | 33
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 2
  Male | 13 | 18 | 31
Region of Enrollment [Number; unit: participants]
  United States | 15 | 18 | 33

OUTCOME MEASURES:

1. Primary Outcome: Total Number of Subjects With Reported Side Effects as Assessed by Dosage Record and Treatment Emergent Symptom Scale (DOTES)
Description: The Dosage Record and Treatment Emergent Symptom Scale (DOTES) provides information on the presence, frequency, and severity of side effects reported during the course of the trial.
Time Frame: 4, 8, and 12 weeks
Population: We analyzed subjects who had follow-up data available.
Measure: Number; unit: participants
Arm/Group | N-Acetyl Cysteine | Sugar Pill
Number analyzed (Participants) | 14 | 15
participants
  Total Number of Subjects with GI adverse Events | 11 | 7
  Constipation | 3 | 2
  Nausea/Vomiting | 6 | 3
  Diarrhea | 3 | 1
  Increased Appetite | 2 | 0
  Decreased Appetite | 2 | 3
  Akathisia | 1 | 0
  Excitement/Agitation | 2 | 3
  Increased Motor Activity | 2 | 3
  Tremor | 0 | 1
  Syncope/Dizziness | 0 | 1
  Depressive Affect | 1 | 0
  Nasal Congestion | 4 | 6
  Increased Salivation | 0 | 2
  Sweating | 0 | 1

2. Primary Outcome: The Clinical Global Rating Scale (CGRS) Improvement Subscale Score
Description: Score range 1-7 (lower score mean more improvement compared to baseline)
Time Frame: 12 weeks
Population: We analyzed subjects who had follow-up data available.
Measure: Mean (Standard Deviation); unit: score (range 1-7)
Arm/Group | N-Acetyl Cysteine | Sugar Pill
Number analyzed (Participants) | 14 | 15
score (range 1-7) | 3.2 (0.9) | 2.9 (1.1)
Statistical Analysis 1: Comparison: N-Acetyl Cysteine vs Sugar Pill; Cohen's d = 0.30; Test type: Superiority or Other; p = 0.449, mixed effects regression models; F= 0.81

3. Primary Outcome: Glutathione (GSH) Levels in Peripheral Blood, Measured by State-of-the-art High-performance Liquid Chromatography (HPLC)
Description: Data not collected. The laboratory was not able to measure Glutathione levels.
Time Frame: 12 weeks
Population: Data not collected.
Arm/Group | N-Acetyl Cysteine | Sugar Pill
Number analyzed (Participants) | 0 | 0

4. Primary Outcome: Irritability Subscale of the Aberrant Behavior Checklist (ABC)
Description: Aberrant Behavior Checklist (ABC) Irritability Subscale Score (range 0-45); higher scores mean higher irritability
Time Frame: baseline and 12 weeks
Population: We analyzed subjects who had follow-up data available.
Measure: Mean (Standard Deviation); unit: Score (range 0-45)
Arm/Group | N-Acetyl Cysteine | Sugar Pill
Number analyzed (Participants) | 14 | 15
Score (range 0-45)
  Baseline ABC-I Score | 16.9 (7.9) | 14.8 (9.6)
  Week 12 ABC-I Score | 7.2 (5.7) | 13.1 (9.9)
Statistical Analysis 1: Comparison: N-Acetyl Cysteine vs Sugar Pill; F values were derived from the interaction of participant group (NAC vs. placebo) and time (week) in mixed effects regression models. Cohen's d was computed based on the standardized mean difference in the change from baseline to week 12; Test type: Superiority or Other; p < .001, Mixed effects regression models — Aberrant Behavior Checklist irritability subscale (F = 6.80; p = <.001; d = .96)

5. Secondary Outcome: The Aberrant Behavior Checklist Total Score (ABC)
Description: Total score was not analyzed since we analyzed the sub scales. Additionally, the authors of the instrument do not recommend analyzing the total score.
Time Frame: 4, 8, and 12 weeks
Population: Measure not analyzed.
Arm/Group | N-Acetyl Cysteine | Sugar Pill
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Social Responsiveness Scale (SRS)
Description: SRS total score (range 0-195); higher scores mean more social impairment
Time Frame: 12 weeks
Population: We analyzed subjects who had follow-up data available.
Measure: Mean (Standard Deviation); unit: SRS total score (range 0-195)
Arm/Group | N-Acetyl Cysteine | Sugar Pill
Number analyzed (Participants) | 14 | 15
SRS total score (range 0-195)
  Baseline SRS Total Score | 111.9 (28.3) | 104.7 (28.1)
  Week 12 SRS Total Score | 93.8 (26.7) | 98.5 (37.8)
Statistical Analysis 1: Comparison: N-Acetyl Cysteine vs Sugar Pill; F-values were derived from the interaction of Participant Group (NAC vs. Placebo) and Time (Week) in mixed effects regression models; Test type: Superiority or Other; p = .141, mixed effects regression models; degrees of freedom were 1, 22

7. Secondary Outcome: Sensory Profile Questionnaire (SPQ)
Time Frame: 12 weeks
Population: Data not collected. Measure not analyzed.
Arm/Group | N-Acetyl Cysteine | Sugar Pill
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Glutathione (GSH) Metabolism Intermediates in Peripheral Blood
Time Frame: 12 weeks
Population: Data not collected. The measure was not analyzed. The lab was not able to measure Glutathione for the study.
Arm/Group | N-Acetyl Cysteine | Sugar Pill
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline and 4, 8 and 12 Weeks
Description: We analyzed all subjects who had follow-up data available.
Arm/Group | N-Acetyl Cysteine | Sugar Pill
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/15
Other Adverse Events (participants affected / at risk) | 13/14 | 14/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | N-Acetyl Cysteine (N=14) | Sugar Pill (N=15)
Constipation (Gastrointestinal disorders) | 3 (3) | 2 (2)
Nausea/Vomiting (Gastrointestinal disorders) | 6 (6) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 3 (3) | 1 (1)
Increased Appetite (Gastrointestinal disorders) | 2 (2) | 0 (0)
Decreased Appetite (Gastrointestinal disorders) | 2 (2) | 3 (3)
Akathisia (General disorders) | 1 (1) | 0 (0)
Excitement/ Agitation (General disorders) | 2 (2) | 3 (3)
Increased Motor Activity (General disorders) | 2 (2) | 3 (3)
Tremor (General disorders) | 0 (0) | 1 (1)
Syncope/Dizziness (General disorders) | 0 (0) | 1 (1)
Depressive Affect (Psychiatric disorders) | 1 (1) | 0 (0)
Nasal Congestion (General disorders) | 4 (4) | 6 (6)
Increased Salivation (General disorders) | 0 (0) | 2 (2)
Sweating (General disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
The sample size was relatively small and the age range was narrow, which limits the generalizability of the findings. Most subjects were taking psychotropic medications and were receiving behavioral interventions.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No